CLINICAL TRIAL: NCT05681988
Title: Early Minimally Invasive Image Guided Endoscopic Evacuation of Intracerebral Haemorrhage (EMINENT-ICH): a Randomized Controlled Trial
Brief Title: Early Minimally Invasive Image Guided Endoscopic Evacuation of Intracerebral Haemorrhage (EMINENT-ICH)
Acronym: EMINENT-ICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); University Hospital, Geneva (Other); Cantonal Hospital of St. Gallen (Other); Ospedale Regionale di Lugano (Other); Centre Hospitalier Universitaire Vaudois (Other); Hôpital du Valais (Other); University Hospital, Zürich (Other); Kantonsspital Winterthur KSW (Other); Insel Gruppe AG, University Hospital Bern (Other); Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-02216; ko22Guzman
Record Dates: First submitted 2022-12-20; First posted 2023-01-12 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Intracerebral Haemorrhage
Keywords: spontaneous supratentorial intracerebral haemorrhage (SSICH); best medical treatment (BMT); surgical hematoma evacuation; conventional craniotomy (CC); early image-guided endoscopic surgery; endoscopic surgery (ES); minimally invasive surgery (MIS); minimally invasive puncture surgery (MIPS); stereotactic aspiration (SA)
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: National multi-centre, two-arm, open labelled randomised controlled trial within the stroke units and stroke centres of the swiss stroke registry in a superiority fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Intervention (Experimental): Early minimally invasive image guided endoscopic hematoma evacuation as an add-on therapy to BMT performed within 24 hours after SSICH symptom onset.
  Interventions: Procedure: Early minimally invasive image guided endoscopic hematoma evacuation; Procedure: Best medical treatment (BMT)
- Control Intervention (Active Comparator): Best medical treatment i.e. active blood pressure control, seizure prophylaxis and care as according to the current guidelines.
  Interventions: Procedure: Best medical treatment (BMT)

INTERVENTIONS:
Procedure: Early minimally invasive image guided endoscopic hematoma evacuation — The intervention group will first receive BMT (as defined below) upon admission and early minimally invasive image guided endoscopic hematoma evacuation as an add-on therapy to BMT. Surgery will be performed within 6-24 hours after SSICH symptom onset. Surgery will be performed in an emergency operating theatre or a hybrid operation theatre equipped with intraoperative CT (in hybrid OR), neuronavigation, and neuro-endoscopy.The position and progress of the trocar towards the hematoma cavity will be monitored with neuro-navigation. The endoscope (LOTTA® system, Karl Storz Endoscopes, Germany; Minop®, BBraun, Tuttlingen, Germany or equivalent) will be inserted into the trocar and tracked using neuro-navigation. Using the pre-planned trajectory, the hematoma will be entered. Using continuous suction and irrigation, the hematoma will be aspirated and/or washed out.
  Arms: Study Intervention
Procedure: Best medical treatment (BMT) — The control group will receive the current gold standard treatment for SSICH according to the guidelines (BMT). This involves strict blood pressure control (SBP<140mmHg), if needed with intravenous or intraarterial blood pressure lowering agents, reversal of anticoagulation if applicable, intensive care surveillance and nursing on a ICU or stroke unit, control of seizures as well as glucose levels as needed and neurointensive monitoring if deemed necessary

SUMMARY:
This is an open-labelled, single centre randomised controlled trial evaluating the efficacy of early minimally invasive image-guided hematoma evacuation in combination with the current best medical treatment compared to best medical treatment alone in improving functional outcome rates at 6 months after initial treatment in patients with spontaneous supratentorial intracerebral haemorrhage.

DETAILED DESCRIPTION:
Spontaneous supratentorial intracerebral haemorrhage (SSICH) is the second most common form of stroke and accounts for approximately 2500 cases in Switzerland annually. The prognosis is very poor with nearly half of the patients dying within one year after haemorrhage. Treatment options for SSICH consist of either the current gold standard, best medical treatment (BMT), or surgical hematoma evacuation. Neither the best medical treatment nor the established surgical mainstay (conventional craniotomy) have shown relevant improvement of survival or functional outcome rates. A minimal invasive approach with early image-guided endoscopic surgery conducted within 24 hours after bleeding onset is therefore proposed. Endoscopic surgery was shown to be safe and effective, however large trials analyzing the benefits of endoscopic surgery are lacking. An earlier, more complete and more rapid hematoma evacuation could improve the functional outcome and mortality rates in affected patients. The primary objective of this two-armed, open-labelled, single centre randomised controlled trial is to show superiority of early minimally invasive image-guided hematoma evacuation additionally to BMT compared to BMT alone in improving functional outcome rates at 6 months in patients with SSICH. The study procedures include 6 visits in total, 4 of them during hospital stay, 2 of them as follow-up visits within the clinical routine. Each visit consists of assessing Glasgow Coma Scale (GCS), modified Rankin Scale (mRS) and National Institute of Health Stroke Scale (NIHSS), three visits include CT scans (before intervention, directly postoperative and during follow up) and blood sampling (before intervention, postoperative and during follow up). Three visits include assessing patient satisfaction and cognition, and two visits include patient quality of life assessments. This study was designed in collaboration with Patient and Public representatives.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous supratentorial intracerebral hemorrhage (SSICH), defined as the sudden occurrence of bleeding into the lobar parenchyma and/or into the basal ganglia and/or thalamus that may extend into the ventricles confirmed by imaging
* SSICH volume ≥20 mL <100 mL
* A focal neurological deficit consisting of either

  * clinically relevant hemiparesis (≥4 motor points on the NIHSS for facial palsy, motoric upper and lower extremities combined)
  * clinically relevant motor or sensory aphasia (≥2 points on the NIHSS)
  * clinically relevant hemi-inattention (formerly neglect, 2 points on the NIHSS)
  * decreased level of consciousness (Glasgow Coma Scale (GCS)≤13)
* Presenting GCS 5 - 15 (in intubated patients GCS assessment will be performed after Rutledge et al. or if impossible, the last pre-intubation GCS will be used)
* Endoscopic hematoma evacuation can be initiated within 24 hours after the patient was last seen well/symptom onset
* Informed consent of patient or appropriate surrogate (for patients without competence)

Exclusion Criteria:

* SSICH due to known or suspected structural abnormality in the brain (e.g. vascular malformation, aneurysm, arteriovenous malformation (AVM), brain tumor) and/or brain trauma and/or hemorrhagic conversion of an ischemic infarction
* Multiple simultaneous intracranial hemorrhages (ICH) (e.g. multifocal ICH, chronic subdural hematoma (cSDH), acute subdural hematoma (aSDH), SAH)
* Infratentorial hemorrhage or midbrain extension/involvement of the hemorrhage
* Coagulation disorder (including anticoagulation) with an international normalized ratio (INR) of >1.5 which cannot be pharmacologically reverted until the planned time of evacuation
* Pregnancy
* Relevant disability prior to SSICH (mRS >2)
* Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments through 180 days (e.g. bilateral fixed dilated pupils)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Good functional outcome, measured by the modified Rankin Scale (mRS) | At 6 months after treatment
  Good functional outcome is defined as a mRS of ≤3 points and will be assessed as binary outcome (yes/no, final value). In this context, a mRS score of 3 points reflects the ability to walk unassisted and care for one's own bodily needs despite being moderately dependent on assistance, while a mRS score of 4 points describes a patient who is not able to walk anymore and needs assistance with all daily activities and thus marks a severe loss of patient autonomy.

SECONDARY OUTCOMES:
Mortality rate | At 6 and 12 months after intervention
  Mortality rate as measured by death of a participant (binary outcome (yes/no)
Change in Quality of Life, assessed by Patient-Reported Outcomes Measurement Information System (PROMIS®) questionnaire | At 3 and 6 months after intervention
  The PROMIS® questionnaire scores can be categorized as: within normal limits, mild, moderate and severe.
Change in Patient cognitive outcome as assessed by the Montreal-Cognitive-Assessment-Test (MOCA® ) | At 3 and 6 months after intervention
  The MOCA assesses: Short term memory. Visuospatial abilities. Executive functions. Attention, concentration and working memory. Language.18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment and less than 10= severe cognitive impairment. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal.
Morbidity rate | At 6 and 12 months after intervention
  The morbidity rate, meaning occurrence of: Ischemic stroke, Recurrent SSICH (defined as any radiologically confirmed increase in hematoma volume postoperative/follow-up that is either asymptomatic or associated with a worsening of the focal-neurological deficit by ≥4 points on the NIHSS and/or a decrease in consciousness by ≥2 points on the GCS), Epileptic seizure, Surgical site infection (intervention group only), Any need for open neurosurgical procedures, Infections (i.e. pneumonia, urinary tract infection), Any other not defined complication that prolongs the hospital stay and/or leads to further treatment not envisaged in the original treatment plan.
Change of focal neurological deficit measured by the National Institute of Health Stroke Scale (NIHSS) | From baseline to 6 months after intervention
  The NIHSS is composed of 11 items. The score for each ability is a number between 0 and 4, 0 being normal functioning and 4 being completely impaired.
Time to intervention | At baseline
  Time to intervention, defined as the period from symptom onset/last seen well to start of surgery (start surgical measures, i.e. positioning of patient) or start of medical treatment (admission of first treatment of BMT) (continuous variable, time to event).
Total time spent on the intensive care unit (ICU)/stroke unit | At 7 days/discharge after intervention
  The total time spent on the intensive care unit (ICU)/stroke unit as a continuous variable from the first admission to the ICU/stroke unit to discharge from ICU/stroke unit
Total time spent in intubation measured in minutes | At 7 days/discharge after intervention
  The total time spent in intubation measured in minutes from the start of intubation to extubation as specified in the anesthesiology report
Proportion of hematoma volume reduction rate (in the intervention group only) | Directly after intervention
  The hematoma volume will be measured on serial cranial computer tomography (cCT) and the difference between the volume of the cCT used for surgery and the cCT directly after surgery will be calculated.
Change in Patient Satisfaction Questionnaire | At 3 and 6 months after intervention
  Patient Satisfaction as assessed by a 5- item survey on a scale of 1-5 (Score (1=worst, 5=best)

CONTACTS AND LOCATIONS:
Overall Officials: Jehuda Soleman, Prof. Dr. med., Principal Investigator — Department of Neurosurgery, University Hospital Basel
Locations (10):
- Switzerland (10):
  - Department of Neurosurgery, University Hospital Basel, Basel
  - University Hospital Bern, Bern
  - Hopitaux Universitare Geneve, Geneva
  - Centre Hopitalier Universitaire Vaudoise, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Ospedale Regionale di Lugano, Lugano
  - Kantonsspital St. Gallen, Sankt Gallen
  - Centre Hopitalier Universitaire du Valais Romand, Sion
  - Kantonsspital Winterthur, Winterthur
  - Universitätsspital Zürich, Zurich

REFERENCES:
- [Background] Hallenberger TJ, Guzman R, Soleman J. Minimally invasive image-guided endoscopic evacuation of intracerebral haemorrhage: How I Do it. Acta Neurochir (Wien). 2023 Jun;165(6):1597-1602. doi: 10.1007/s00701-022-05326-3. Epub 2022 Aug 5. PMID 35930078
- [Derived] Hallenberger TJ, Fischer U, Ghosh N, Kuhle J, Guzman R, Bonati LH, Soleman J. Early minimally invasive image-guided eNdoscopic evacuation of iNTracerebral hemorrhage: a phase II pilot trial. Front Neurol. 2024 Nov 19;15:1484255. doi: 10.3389/fneur.2024.1484255. eCollection 2024. PMID 39628893
- [Derived] Hallenberger TJ, Fischer U, Bonati LH, Dutilh G, Mucklow R, Vogt AS, Boeni-Eckstein C, Cardia A, Schubert GA, Bijlenga P, Messerer M, Raabe A, Akeret K, Zweifel C, Kuhle J, Alfieri A, Fournier JY, Fandino J, Hostettler IC, Schneider UC, Guzman R, Soleman J. Early minimally invasive image-guided endoscopic evacuation of intracerebral hemorrhage (EMINENT-ICH): a randomized controlled trial. Trials. 2024 Oct 18;25(1):692. doi: 10.1186/s13063-024-08534-7. PMID 39425219
- See also: Publication with PMID35930078: "Minimally invasive image-guided endoscopic evacuation of intracerebral haemorrhage: How I Do it" — https://link.springer.com/article/10.1007/s00701-022-05326-3